CLINICAL TRIAL: NCT05843799
Title: A Phase I, Single-center, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety and Tolerability of ILB-202 Administered Intravenously As Single Ascending Doses to Healthy Participants
Brief Title: A Study to Evaluate the Safety and Tolerability of ILB-202
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ILIAS Biologics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ILB-202-001
Record Dates: First submitted 2023-03-31; First posted 2023-05-06 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ILB-202 (Experimental): ILB-202 exosome with Clinical grade normal saline (0.9% sodium chloride for intravenous injection)
  Interventions: Drug: ILB-202
- Placebo (Placebo Comparator): Clinical grade normal saline (0.9% sodium chloride for intravenous injection)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ILB-202 — Single i.v. infusion
  Arms: ILB-202
Drug: Placebo — Single i.v. infusion
  Arms: Placebo

SUMMARY:
This is a Phase I, Single-center, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety and Tolerability of ILB-202 Administered Intravenously as Single Ascending Doses to Healthy Participants. Male or female subjects aged 18 to 50 years (inclusive) who fulfill the inclusion/exclusion criteria will be enrolled in this study.

DETAILED DESCRIPTION:
ILB-202 is an engineered exosome loaded with super-repressor IκBα. This is Phase I, Single-center, Randomized, Double-blind, Placebo-controlled Study.

Healthy volunteers, 18-55 years of age, selected from healthy participants fulfilling the inclusion/exclusion criteria.

18 subjects will participate in the study. Doses of investigational product (IP) will be administered intravenously on Day 1. During the Screening Period (within the 28 days) each subject will be assessed for eligibility. Each subject must sign and date an informed consent form (ICF) prior to undergoing any study-related procedures.

All dosed subject samples will be analyzed and their data will be included in the final study report.

ELIGIBILITY:
Inclusion Criteria:

* Must have given written informed consent and must be able to understand the full nature and purpose of the trial.
* Aged 18 to 55 years of age (inclusive).
* A body mass index (BMI) of ≥ 18.0 and ≤ 30.0 kg/m2 .
* Medically healthy male or female volunteers, without clinically significant abnormalities.
* Conventional 12-lead ECG recording in triplicate consistent with normal cardiac conduction and function.
* Must be of non-child-bearing potential, or must be on a suitable birth control method.

Exclusion Criteria:

* History or evidence of any clinically significant condition and/or other major disease or malignancy.
* History of drug allergies and drug or alcohol abuse .
* Clinically significant abnormalities in the physical examination, vital signs, ECG or clinical laboratory tests.
* Exposure to any prescription medications or, administered over the counter drugs, dietary supplements, or herbal remedies, within 14 days or 5 half-lives, prior to dosing.
* Received treatment with immune-suppressive or immune-modulative medication within 90 days prior to dosing.
* Exposure to biologics within 6 months prior to dosing.
* Participation in another clinical trial within 30 days (or 6 months for biologics) prior to dosing.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2023-05-16 (Actual); Primary Completion 2023-10-04 (Actual); Study Completion 2023-10-04 (Actual)

PRIMARY OUTCOMES:
Incidence, severity and relationship to study treatment of Adverse Events(AEs) | Day 1 (administration) through Day 8
  Number of participants with adverse events as assessed by Common Terminology Criteria for Adverse Events(CTCAE) v5.0
Concomitant medication usage | Day 1 (administration) through Day 8
  Number of participants with new(additional) treatment
Specific Parameter Change from Baseline to End of Study | Day 1 (administration) through Day 8
  Number of participants with clinically significant changes in
  * body weight
  * vital signs
  * Electrocardiogram(ECG) parameters
  * clinical laboratory parameters

OTHER OUTCOMES:
Rate of immune cell activation markers | Day 1 (administration) through Day 3
  * Rate of T cell
  * Rate of B cell
  * Rate of Natural Killer(NK) cell
Component Rates in Distinct Blood Specimens | Day 1 (administration) through Day 2
  * Components rate of plasma
  * Components rate of Red blood cell (RBC)-lysed whole blood
  * Components rate of Peripheral blood mononuclear cells (PBMCs)

CONTACTS AND LOCATIONS:
Locations (1):
- Adelaide, Adelaide, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hyun S, Choi H, Sub Y, Hong D, Ahn SH, Choi K, Ryu S, Kim Y, Park C, Gee HY, Choi C. Safety and Anti-Inflammatory Effects of Engineered Extracellular Vesicles (ILB-202) for NF-kappaB Inhibition: A Double-Blind, Randomized, Placebo-Controlled Phase 1 Trial. J Extracell Vesicles. 2025 Sep;14(9):e70141. doi: 10.1002/jev2.70141. PMID 41002119